CLINICAL TRIAL: NCT03712475
Title: A Randomized, Single-dose, Parallel-group Study to Evaluate the Pharmacokinetic Profiles of Two Formulation of Pregabalin in Healthy Volunteers Under Fasting Conditions
Brief Title: Pharmacokinetics of Two Formulation of Pregabalin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RJH3001-01
Record Dates: First submitted 2018-10-08; First posted 2018-10-19 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Peripheral Neuropathy; Fibromyalgia; Partial Seizure Disorder
Keywords: Pharmacokinetic
MeSH Terms: conditions — Fibromyalgia; Epilepsies, Partial | interventions — Pregabalin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phudialin Hard Capsules (Experimental): Phudialin Hard Capsules Dosing Regimen: Single dosing
  Interventions: Drug: Pregabalin
- Lyrica Hard Capsule (Active Comparator): Lyrica Hard Capsule Dosing Regimen: Single dosing
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — pharmacokinetic study under fasting conditions

SUMMARY:
A Randomized, Single-Dose, Parallel-Group Study to Evaluate the Pharmacokinetic Profiles of Two Formulations of Pregabalin after Oral Administration in Healthy Volunteers under Fasting Conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects between 20-45 years of age.
2. Body weight within 80-120% of ideal body weight.

   * Ideal body weight (kg) = [height (cm) - 80] *0.7 for male subjects
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in chest x-ray and electrocardiogram results within six months prior to study drug dosing.
   * no particular clinical significance in general disease history within two months prior to study drug dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes Serum Glutamic Oxaloacetic Transaminase (SGOT, same as AST), Serum Glutamic Pyruvic Transaminase (SGPT, same as ALT), Gamma-Glutamyl-Transpeptidase (γ-GT), alkaline phosphatase, total bilirubin, albumin, glucose, Blood Urea Nitrogen(BUN), uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes power of hydrogen (pH), blood, glucose, ketones, bilirubin and protein.
7. Male subjects willing to use a condom during any sexual contact with females of reproductive potential for up to 10 weeks after study drug dosing.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the investigator).
2. A clinically significant illness or surgery within four weeks prior to study drug dosing (as determined by the investigator).
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime as judged by the investigator.
6. History of alcohol addiction or abuse within last five years as judged by the investigator.
7. History of allergic response(s) to pregabalin or any other related drugs.
8. Evidence of chronic or acute infectious diseases.
9. Positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to study drug dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
11. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to study drug dosing.
12. Use of any investigational drug within four weeks prior to study drug dosing.
13. Donating more than 250 mL of blood within two months prior to study drug dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to study drug dosing.
14. Any other medical reason as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration (AUC) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours
Peak Drug Concentration (Cmax) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours
Elimination half-life (T1/2) | Time Frame: Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours
Area under the (first) moment plasma concentration-time curve (AUMC) | Plasma sample: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 and 36 hours

SECONDARY OUTCOMES:
Adverse events | Within 8 weeks prior to the study, subjects were screened for their eligibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan